CLINICAL TRIAL: NCT01804374
Title: A Phase II, Open Label, Non-randomized Study of Second or Third Line Treatment With the Combination of Sorafenib and Everolimus in Patients Affected by Relapsed and Non-resectable High-grade Osteosarcoma
Brief Title: Phase II Open Label, Non-randomized Study of Sorafenib and Everolimus in Relapsed and Non-resectable Osteosarcoma
Acronym: SERIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SERIO
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Osteosarcoma; Relapsed Osteosarcoma
Keywords: osteosarcoma; sorafenib; everolimus; sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma | interventions — Sorafenib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib and everolimus (Experimental): This is an open label study: all patients will be treated with sorafenib 400 mg twice a day in combination with everolimus 5mg per day
  Interventions: Drug: Sorafenib; Drug: Everolimus

INTERVENTIONS:
Drug: Sorafenib — Sorafenib tablet 200 milligrams packed in bottle containing 140 tablets. Sorafenib will be administered orally twice daily at the same time every day. Two 200 mg tablets will be taken either one hour before or two hours after a meal followed by a glass of water in the morning and in the evening. In general, patient should have a low to moderate fat meal. Patients will receive Sorafenib until progression, toxicity, withdrawal of informed consent or clinical investigator decision
  Other Names: BAY 43-9006; Nexavar
Drug: Everolimus — Everolimus is formulated in tablets of 2.5 or 5 mg strength, blister-packed under aluminum foil in units of 10 tablets. Everolimus will be administered orally once daily at the same time every day immediately after a meal, as a single dose of 5 mg. Patients should have a low-fat breakfast. After this light meal, study medication of Everolimus is to be taken. The tablets of Everolimus should not be chewed or crushed. Patients will receive Everolimus until progression, toxicity, withdrawal of informed consent or clinical investigator decision
  Other Names: RAD001; Afinitor; Certican

SUMMARY:
This is a trial for patients affected by metastatic or relapsed osteosarcoma which progressed after first or further line treatments. In this trial, all patients will be treated until progression or unacceptable toxicity with sorafenib and everolimus. The treatment with sorafenib and everolimus aimed to obtain a 50% rate of patients free from further progression of the disease after 6 months from study entry.

DETAILED DESCRIPTION:
Patients affected by metastatic or relapsed osteosarcoma which progressed after first or further line treatments still have a poor outcome. Standard chemotherapy has limited activity in these patients.

In a previous study in patient affected by relapsed unresectable osteosarcoma, sorafenib alone demonstrated promising activity. In the preclinical setting, everolimus was able to improve the activity of sorafenib. Sorafenib and everolimus, by hitting crucial pathways which are essential for osteosarcoma cell proliferation and survival, with an entirely different approach aimed to overcome the resistance to standard chemotherapy showed by relapsed osteosarcoma. In this trial, all patients will be treated with sorafenib and everolimus at the dosage of 800 mg and 5 mg per day, respectively. Both drugs have to be taken orally. The treatment will be continued until progression or unacceptable toxicities. The objective of the present trial is to obtain a 50% rate of patients alive and free from progression of their disease 6 months after trial enrolment. The disease will be evaluated every 2 months with a CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented and not surgically resectable or metastatic high-grade osteosarcoma which progressed after first or second line treatments for relapsing disease
* Measurable disease as defined by RECIST criteria vs. 1.1 (bone lesions are allowed). Baseline evaluations must be completed within 28 days prior to enrollment
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1. ECOG PS 2 patients are eligible if the PS 2 depends solely on orthopedic problems
* Estimated life expectancy of at least 3months
* Age≥18 years
* Adequate bone marrow, liver and renal function: Hemoglobin>9.0g/dl, Absolute neutrophil count>1,500/mm3, Platelet>100,000/μl Total bilirubin<1.5 times the upper limit of normal (ULN), ALT and AST<2.5xULN (<5xULN for patients with liver involvement of their cancer), PT-INR/PTT<1.5xULN, Serum creatinine<2xULN
* Written informed consent

Exclusion Criteria:

* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Patients with any severe and/or uncontrolled medical conditions such as unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6months, serious uncontrolled cardiac arrhythmia, uncontrolled hyperlipidemia, active or uncontrolled severe infection, cirrhosis, chronic or persistent active hepatitis or severely impaired lung function.
* History of HIV infection and active clinically serious infections (>grade 2 according to NCI-CTCAE vs. 4.0)
* Symptomatic metastatic brain or meningeal tumors (unless the patient is >6months from definitive therapy, has a negative imaging study within 4weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
* Patients with seizure disorders requiring medication
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7days of the start of treatment. Both men and women must use adequate barrier birth control measures during the course of the trial and 8weeks after last dose of study drug
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Patients unable to swallow oral medications
* Uncontrolled diabetes (fasting glucose>2xULN)
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent (except corticosteroids with a daily dosage equivalent to prednisone ≤20mg for adrenal insufficiency). Patients receiving corticosteroids must be on a stable dose for ≥4weeks prior to the first dose of Everolimus. Topical or inhaled corticosteroids are permitted
* Patients with a history of another malignancy within 5years prior to study entry, except curatively treated non-melanotic skin cancer or in-situ cervical cancer skin or other solid tumors curatively treated with no evidence of disease for ≥3years. Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Anticancer chemotherapy or immunotherapy during the study or within 4weeks of study entry
* Radiotherapy during study or within 3weeks of start of study drug. (Palliative radiotherapy will be allowed)
* Major surgery within 4weeks of start of study
* Investigational drug therapy outside of this trial during or within 4weeks of study entry
* Prior exposure to the study drugs or their analogues
* Patients with known hypersensitivity to sorafenib, everolimus or other rapamycin analogs, or to its excipients
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* A history of noncompliance to medical regimens or inability or unwillingness to return for scheduled visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival rate at 6 months | 6 months from registration into the study
  Progression Free Survival rate at 6 months refers to the rate of patients alive and free from progression of the disease at 6 months from registration into the study. Disease will be assessed every 8 weeks up to 2 years until progression or death whichever came first.

SECONDARY OUTCOMES:
progression free survival | From randomization until progression or death whichever came first up to 2 years
  Progression Free Survival (PFS) refers to the time from registration into the study to the date of progressive disease or death whichever came first assessed every 8 weeks up to 2 years. In the absence of progression, time will be censored at the date of last tumor assessment or follow-up
overall survival | From randomization until death followed up to 5 years
  Overall survival (OS) is the time interval between date of registration into study and the date of death. For alive patients, time will be censored at the date of last follow-up.
Overall response rate | From randomization until progression or death whichever came first up to 2 years
  Overall response rate refers to the rate of patients with complete, partial or minimal responses (defined as shrinkage of target lesions between 10 and 30%) according to RECIST 1.1. Disease will be assessed every 8 weeks up to 2 years.
Duration of response | calculated from date of first assessement of non-progression until progression or death whichever came first up to 2 years
  Duration of response refers to the time from the date of the first assessement of non-progression to the date of progressive disease or death. Disease will be assessed every 8 weeks up to 2 years until progression or death whichever came first. In the absence of progression time will be censored at the date of last tumor assessment or follow-up.
Non-dimensional pattern of response | calculated from randomization until progression or death whichever came first up to 2 years
  Non-dimensional pattern of response refers to the evaluation of any consistent variation in radio metabolic diagnostic test (i.e. PET or Bone scan) and/or changes in signal intensity, contrast uptake/enhancement and tumor density at CT/MRI according to Modified Response Criteria (MRC). From this point of view, patients will be considered in response if there has been an objective response or at least ONE of the following criteria are met:
  1. An unequivocal reduction in tumor density at CT scan;
  2. An unequivocal reduction in signal intensity and/or contrast enhancement at MRI;
  3. An unequivocal reduction in SUV at PET scan;
  4. An unequivocal reduction in bone scan uptake.
  Disease will be assessed every 8 weeks up to 2 years until progression or death whichever came first.
clinical benefit | evaluated at each visit from randomizzation until progression or death whichever came first up to 2 years
  Clinical Benefit will be prospectively evaluated by means of Pain and Analgesic Scale recording of analgesic consume and as lack of progression of disease at six months.
Safety | assessed at each visit from randomizzation until 28 days after the last dose of study treatment assumption up to 2 years
  Safety will be captured by recording: physical examinations, vital signs, performance status/body weight; blood tests and chemistry tests; intensity and severity of adverse events, use of analgesic medication at each visit until 28 days after last dose of study treatment assumption up to 2 years. Adverse events will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

OTHER OUTCOMES:
Expression of MAPKs pathway, VEGFR, PDGFR, Ezrin/Moesin and mTOR pathway (pS6 expression) | as soon as tissue samples are available or within 2 months from subject study entry
  Immunohistochemical evaluation of the expression of MAPKs pathway, VEGFR, PDGFR, Ezrin/Moesin and mTOR pathway (pS6 expression)on tissue samples from primary or metastatic tumors.
Correlation between oncogenes/metabolic pathways and clinical outcome parameters | at the time of first survival analysis performed at least 6 months after last subject registration
  Correlation of both primary and secondary objectives with the expression of the following oncogenes/metabolic pathways: MAPKs, VEGFR, PDGFR, Ezrin/Moesin and mTOR pathway (pS6 expression)
Predictive and prognostic role of serum lactate dehydrogenase and serum alkaline phosphatase | at the time of first survival analysis performed at least 6 months after last subject registration
  Serum samples for evaluation of levels of lactate dehydrogenase (LDH) and alkaline phosphatase (ALP) will be collected at each visit until progression or death whichever came first up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Aglietta, MD, Principal Investigator — IRCC Candiolo; Giovanni Grignani, MD, Study Director — IRCC Candiolo; Piero Picci, MD, Study Chair — Italian Sarcoma Group
Locations (1):
- Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino, Italy

REFERENCES:
- [Derived] Grignani G, Palmerini E, Ferraresi V, D'Ambrosio L, Bertulli R, Asaftei SD, Tamburini A, Pignochino Y, Sangiolo D, Marchesi E, Capozzi F, Biagini R, Gambarotti M, Fagioli F, Casali PG, Picci P, Ferrari S, Aglietta M; Italian Sarcoma Group. Sorafenib and everolimus for patients with unresectable high-grade osteosarcoma progressing after standard treatment: a non-randomised phase 2 clinical trial. Lancet Oncol. 2015 Jan;16(1):98-107. doi: 10.1016/S1470-2045(14)71136-2. Epub 2014 Dec 11. PMID 25498219